CLINICAL TRIAL: NCT03205748
Title: Evaluation of Different Etiologies of Obscure Ascites: Clinical, Laboratory, and Laparoscopic Study.
Brief Title: Evaluation of Different Etiologies of Obscure Ascites
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: OA
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ascites refers to fluid that accumulates within the peritoneal cavity. Although ascites is most commonly observed in patients with cirrhosis and resulting portal hypertension (approximately 85% of cases), 7% to 10% of patients with ascites develop secondary to a malignancy

ELIGIBILITY:
Inclusion Criteria:

* Patients with ascites
* serum ascites albumin gradient >1.1.

Exclusion Criteria:

* ascitic fluid serum ascites albumin gradient <1.1.
* Haemorrgaic ascites;
* chylous ascites

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients will be recruited from Departments of Internal Medicine, Assiut university tertiary hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with malignant ascites | 1 month
  according to laboratory and clinical criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt